CLINICAL TRIAL: NCT01388543
Title: Genetic-determinants of Protease Inhibitor Pharmacology
Brief Title: Genetics and HIV-1 Protease Inhibitors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 06-0428; R03AI068438 (NIH); BMSV-338 (Other Grant/Funding Number: Bristol-Myers Squibb)
Record Dates: First submitted 2011-06-28; First posted 2011-07-06 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: HIV
Keywords: Pharmacokinetics; Clinical Pharmacology; Pharmacogenomics; HIV
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYP3A5 Expressors (Active Comparator): A pre-screening genetic test determines CYP3A5 expressor status
  Interventions: Drug: Atazanavir
- CYP3A5 Non-expressors (Active Comparator): A pre-screening genetic test determines CYP3A5 non-expressor status
  Interventions: Drug: Atazanavir

INTERVENTIONS:
Drug: Atazanavir — Atazanavir 400mg once daily for 7 days followed by atazanavir 300mg plus ritonavir 100mg for 7 days
  Other Names: Reyataz; Norvir

SUMMARY:
This study evaluated the blood levels of atazanavir according to a genetic makeup for CYP3A5 (cytochrome P450 3A5, an enzyme that metabolizes atazanavir). The hypothesis was that people with a slow-metabolizing genotype would have higher blood levels of atazanavir compared to people with the normal metabolizing genotype.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years
* Negative HIV screening antibody test
* CYP3A5 expressor status, race, and sex fit an enrollment opening.

Exclusion Criteria:

* Pregnant or breast-feeding
* Medical history of

  * hepatitis B or C,
  * autoimmune disease,
  * active malignancy,
  * kidney disease including nephrolithiasis
* Organ dysfunction manifested by

  * liver transaminases or
  * serum creatinine >1.25 times the upper limit of normal, or
  * any comprehensive metabolic test (except asymptomatic unconjugated hyperbilirubinemia), blood count, or lipid value > Grade I according to Division of AIDS (DAIDS) adverse drug event grading system (appendix).
* Medical history of arrhythmias (including atrial fibrillation, atrioventricular block, and/or pacemaker)
* Any QT interval abnormalities or other congenital arrhythmia syndromes on ECG or

  * Any ECG abnormality that in the opinion of the investigators would preclude entry into the study.
* Medical history of any serious heart condition including:

  * congestive heart failure,
  * myopathies,
  * coronary artery disease, or
  * unexplained syncope.
* Medical history of bleeding disorders (i.e., hemophilia)
* Hyperlipidemia
* Any prescription, herbal, recreational, or over-the-counter medication contraindicated with ritonavir or atazanavir including:

  * substrates/inhibitors/inducers of CYP3A/P-gp,
  * cardio-active medication, or
  * medications that alter the acid in the stomach. The study investigators will review each concurrent medication on a case-by-case basis.
* Inability to refrain from grapefruit or grapefruit juice during the study.
* Investigational drugs within the last 30 days.
* Active alcohol / recreational drug abuse,
* Inability to give informed consent.
* A body mass index below 18.5 or above 34.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Anderson, PharmD, Principal Investigator — University of Colorado Denver and Health Sciences Center
Locations (1):
- University of Colorado Denver and Health Sciences Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- [Result] Anderson PL, Aquilante CL, Gardner EM, Predhomme J, McDaneld P, Bushman LR, Zheng JH, Ray M, MaWhinney S. Atazanavir pharmacokinetics in genetically determined CYP3A5 expressors versus non-expressors. J Antimicrob Chemother. 2009 Nov;64(5):1071-9. doi: 10.1093/jac/dkp317. Epub 2009 Aug 26. PMID 19710077
- [Result] Wempe MF, Anderson PL. Atazanavir metabolism according to CYP3A5 status: an in vitro-in vivo assessment. Drug Metab Dispos. 2011 Mar;39(3):522-7. doi: 10.1124/dmd.110.036178. Epub 2010 Dec 9. PMID 21148251
- [Result] Kile DA, MaWhinney S, Aquilante CL, Rower JE, Castillo-Mancilla JR, Anderson PL. A population pharmacokinetic-pharmacogenetic analysis of atazanavir. AIDS Res Hum Retroviruses. 2012 Oct;28(10):1227-34. doi: 10.1089/aid.2011.0378. Epub 2012 Apr 20. PMID 22394315

RESULTS

PARTICIPANT FLOW:
Period: Day 7, Primary End Point
Arm/Group | CYP3A5 Expressors | CYP3A5 Non-expressors
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Day 14
Arm/Group | CYP3A5 Expressors | CYP3A5 Non-expressors
Started | 15 | 16
Completed | 14 | 12
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYP3A5 Expressors | CYP3A5 Non-expressors | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 8 | 7 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 7 | 6 | 13
  Hispanic | 3 | 1 | 4
  Asian | 1 | 0 | 1
  Caucasian | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Day 7 Atazanavir Oral Clearance
Description: Measure atazanavir oral clearance in genetically-determined CYP3A5 expressors versus CYP3A5 non-expressors
Time Frame: Day 7
Measure: Geometric Mean (95% Confidence Interval); unit: L/h/kg
Arm/Group | CYP3A5 Expressors | CYP3A5 Non-expressors
Number analyzed (Participants) | 15 | 16
L/h/kg | .25 [.2 to .30] | .18 [.15 to .22]

ADVERSE EVENTS:
Time Frame: Time of consenting to study exit (Day 14 or earlier)
Description: AEs were graded per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, V1.0 Aug 2009 (US Dept HHS, NIH, NIAID) Available from: http://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf
Groups:
- CYP3A5 Expressor; CYP3A5 Non-expressors: A pre-screening genetic test determines CYP3A5 expressor status
  Atazanavir: Atazanavir 400mg once daily for 7 days followed by atazanavir 300mg plus ritonavir 100mg for 7 days
Arm/Group | CYP3A5 Expressor | CYP3A5 Non-expressors
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 1/15 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CYP3A5 Expressor (N=15) | CYP3A5 Non-expressors (N=16)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Abnormal Lab- albumin (Hepatobiliary disorders) | 0 | 1
Unspecified viral syndrome-not study related (General disorders) | 0 | 1
Abnormal Lab- Aspartate transaminase (AST) (Hepatobiliary disorders) | 0 | 1
Abnormal Lab- Amylase (Endocrine disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No